CLINICAL TRIAL: NCT06497946
Title: Effects of the SlimTrack® Platform on Diet Adherence, Body Weight Variation, Anthropometric Variables and Arterial Stiffness in Postmenopausal Women: Pilot Study
Brief Title: Effects of SlimTrack® Platform on Diet Adherence, Anthropometry and Arterial Stiffness in Postmenopausal Women
Acronym: SlimTrack
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Clauda Fetter, Doctor, Instituto de Cardiologia do Rio Grande do Sul
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 6092-23
Record Dates: First submitted 2024-06-13; First posted 2024-07-12 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Menopause; Obesity; Overweight
Keywords: Obesity; Menopause; Weight Loss; Digital Platform; Exercises; Eating Behavior
MeSH Terms: conditions — Obesity; Overweight; Weight Loss; Motor Activity; Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SlimTrack (Active Comparator): Use of the SlimTrack Plataform
  Interventions: Behavioral: SlimTrack Plataform
- SlimTrack + Diet Prescription (Active Comparator): Use of the SlimTrack Plataform + diet prescription
  Interventions: Behavioral: SlimTrack Plataform; Behavioral: Diet prescription
- Diet Prescription (Active Comparator): Use of Diet Prescription
  Interventions: Behavioral: Diet prescription
- Controll (No Intervention): Tips for health with delivery of graphic material

INTERVENTIONS:
Behavioral: SlimTrack Plataform — SlimTrack Plataform requests log in and includes anthropometric data of participants, besides answers about questionaires and other tasks in online content available
  Arms: SlimTrack; SlimTrack + Diet Prescription
Behavioral: Diet prescription — Nutrition Professional evaluates diet habits and prescribes a reeducation method in order to fulfill better behavior towards food intake
  Arms: Diet Prescription; SlimTrack + Diet Prescription

SUMMARY:
Introduction:The weight gain expected in the postmenopausal period has deleterious effects on the physical and mental health of the female population. Management of this situation strongly recommends regular exercise, behavioral and psychological interventions and dietary control. Activities of this nature can be carried out online. The SlimTrack Platform is an interactive digital platform for management and treatment of overweight and obesity in Non-Dietary Weight Loss basis. The first phase consisting of 3 stages of 7 days (total 21 days) presents tools to deal with thoughts and emotions, in addition to offering a series of physical activities that promote body self-awareness and movement needs. Therefore, this study aims to evaluate the effects of this MVP on adherence to the diet, body weight variation, anthropometric variables and arterial stiffness in postmenopausal women, in addition to verifying the accuracy of self-reported measurements on the platform. Methods:Randomized clinical trial will recruit overweight and obese volunteers to evaluate body weight variation, anthropometric variables and arterial stiffness (oscillometric method, obtaining central arterial pressure indices, pulse wave velocity (large artery stiffness) and Aix 75 to identify stiffness of small arteries). Patients will be randomized to the following interventions: Diet, SlimTrack Platform, Diet + SlimTrack Platform and Control. The interventions will have in-person assistance once a week. The data obtained will be analyzed by intention to treat and presented as means (M) ± standard deviation (SD). They will be tested for normality using the Shapiro Wilk test. The differences between interventions will be made through GEE. Correlations between variables will be obtained using Pearson Correlations for parametric data and Spearman Correlations for non-parametric data, with a significance level of p < 0.05. Expected results:Results are expected that point to the effectiveness of non-dietary support (SlimTrack Platform) in both diet adherence and body weight reduction. Furthermore, through comparisons between groups, it will be possible to elucidate the influences of weight reduction, diet and physical activity levels on arterial stiffness.

DETAILED DESCRIPTION:
Obesity is a chronic and multifactorial disease, physiologically characterized by excessive storage of body fat, which may have as a risk factor certain social reasons, lifestyle, inappropriate food consumption, extremely restrictive diets, poor relationship with food, low levels of physical activity, among other aspects. (two) In Brazil, it is estimated that 6 in 10 Brazilians are overweight, which represents 96 million overweight people in the country. Furthermore, according to the World Obesity Federation, by the year 2035, 1 in 4 people (almost two billion) will live with obesity (BMI above 30 kg/m2). Therefore, obesity is the second most important risk factor for the global burden of chronic non-communicable diseases (NCDs), such as cardiovascular diseases , high blood pressure, diabetes, colon, rectum, breast cancer and cirrhosis. However, absence from work, psychological disorders, low self-esteem and social isolation require both a physical and psychological treatment perspective.

A population widely susceptible to weight gain are postmenopausal women. In a physiological context, postmenopause is the last phase of the climacteric period, the reproductive to non-reproductive period, beginning 12 months after the woman's last menstruation, and ending, on average, at 65 years of age. Evidence indicates that 50% of the female population, at this time, has metabolic syndrome, a strong tendency to accumulate visceral abdominal adiposity, seen by an increased abdominal circumference, changes in bone metabolism and greater susceptibility to chronic non-communicable diseases. Among the chronic diseases that develop during menopause are those related to the heart, with high blood pressure, diabetes and coronary disease being the protagonists of this unfavorable scenario, a fact already evidenced by some recent studies that point to women in menopause with a higher prevalence of central arterial stiffness.

Arterial stiffness is the mechanical distension stress induced by anterograde and retrograde systolic waves, which reduces the thickness and fragments elastin fibers, replaced by collagen and protein matrix, with less capacity to dampen pulse wave pressures, increasing the stiffness of the arterial walls and the speed of anterograde and retrograde (or reflex) pulse waves.

Arterial stiffness is assessed using Pulse Wave Velocity (PWV), an important marker of central artery stiffness, considered an early predictor of risk for hypertension and CVD, when PWV > 10 m/s. For every 1 m/s increase in PWV, there is an increase in the risk of cardiovascular death, cardiovascular events and death from all causes of around 14-15%.

A meta-analysis has already demonstrated that reducing body weight (average of 8% of initial body weight), achieved through diet and lifestyle changes, improved PWV. Both diet and regular exercise have an effect on PWV. reduction in PWV as a consequence of weight reduction, and reducing >7% of initial body weight has a more robust effect.

Therefore, the management of body weight during menopause, as well as other aspects of women's health, requires a broad spectrum of transdisciplinary action, with dietary and non-dietary interventions as psychological support and encouragement for a more active life. In this context, new technologies represent a comprehensive and accessible alternative for the use of multidisciplinary tools in body weight management, since technological advances have increasingly provided non-invasive methods for health management.

Therefore, the SlimTrack platform presents tools that help both in facing thoughts and emotions that are harmful to long-term weight loss, and with physical activities that promote body self-awareness, meeting the needs of physical activity, and dietary guidelines, contributing to a change in Lifestyle. At this moment, the platform is in the development process through a notice Call CNPq/SEMPI/MCTI nº 021/2021 - RHAE Program - Line 2 - Start-Ups, Process: 424509/2021-0 Creation of an interactive digital platform for the management and treatment of overweight and obesity - Non-Dietary Weight Loss (END), coordinated by Dr. Cláudia Fetter and Dr. Juliana Bertoletti. The first phase or MVP ( minimum viable product ) is made up of 3 stages of 7 days (total 21 days), is in the finalization phase to be made available to the public, scheduled for October 2023. More information about the platform at the link: https://docs.google.com/document/d/1imApA0fw1f5oqDIvegEY0X3yaE3xRxl2UkERZH_P-yA/edit?usp=sharing

Therefore, in view of the above, as well as the current health scenario and its demands, especially regarding obesity and risk factors associated with health, this project intends to evaluate the effects of the SlimTrack ® Platform on adherence to the diet, variation body weight, anthropometric variables and arterial stiffness in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria

* Menopause
* Overweight
* Obesity
* Sedentary lifestyle

Exclusion Criteria:

* Use of hormone therapy
* Use of pharmacologial pshychiatric medication
* Recent surgery (six months)
* Recent (six months) cardiardiovascular events (myocardial infarction, stroke)
* Adherence to diet in the last six months
* Attending to psychoterapeutic proccess

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cis Women
Enrollment: 64 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Arterial Stiffness (m/s) | Up to 21 days
  Pulse Wave Velocity by oscilometric method, aimed to be decreased at post intervention assessment

SECONDARY OUTCOMES:
Anthropometric Measures (cm) | Up to 21 days
  Abdominal circumference aimed to be decreased at post intervention assessment
Physical Activity Levels | Up to 21 days
  Inventary of Physical Activity Questionnaire (IPAQ) short version aimed to be increased at post intervention assessment
Adherence to Diet | Up to 21 days
  Food Intake Questionnaire (WebDiet) aimed to be increased at post intervention assessment

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Ms Poester, Graduated, Study Director — Instituto de Cardiologia RS
Locations (1):
- Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No